CLINICAL TRIAL: NCT02887352
Title: French Adaptation of the CCST (California Card Sorting Task). Comparison of 3 Packages to CCST With Multiple Sclerosis (MS) Patients
Brief Title: French Adaptation of the California Card Sorting Task (CCST) in Multiple Sclerosis
Acronym: E3C-DIFSEP
Status: Completed | Type: Observational
Sponsor: Fondation Ophtalmologique Adolphe de Rothschild (Network)
Responsible Party: Sponsor
Other Study IDs: OGT_2014-1
Record Dates: First submitted 2016-08-25; First posted 2016-09-02 (Estimated); Last update posted 2021-06-14 (Actual); Status verified 2021-06

CONDITIONS: Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional

INTERVENTIONS:
Other: assessment of problem-solving ability

SUMMARY:
Cognitive impairment affects up to 65% of multiple sclerosis (MS) subjects, especially executive functions. The California Card Sorting Task (CCST) assesses specific components of problem-solving ability. There is currently no French version of this test. Reims neurological department in collaboration with Rothschild Foundation has developed a French adaptation of CCST. This version includes three cards packages with two alternate forms to control practice effects (test-retest). In order to assess "test-retest reliability" we have to verify the comparability of the three cards packages within one session in MS patients.

ELIGIBILITY:
Inclusion Criteria:

* Multiple Sclerosis patients
* age > 18 years old

Exclusion Criteria:

* Montreal Cognitive Assessment (MOCA) ≤20
* psychiatric disease
* no proficiency in the French language
* opposition to participate in the study
* no medical insurance coverage

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: multiple sclerosis patients
Sampling Method: Non-Probability Sample
Enrollment: 48 (Actual)
Dates: Start 2014-03 (Actual); Primary Completion 2020-01 (Actual); Study Completion 2020-01 (Actual)

PRIMARY OUTCOMES:
CCST Test score | baseline
  comparison of the scores of the three versions of the test

CONTACTS AND LOCATIONS:
Overall Officials: Anne-Claire VIRET, Study Director — Fondation OPH A de Rothschild; Olivier GOUT, MD, Principal Investigator — Fondation OPH A de Rothschild
Locations (1):
- Fondation Ophtalmologique Adolphe de Rothschild, Paris, France